CLINICAL TRIAL: NCT03570138
Title: Efficacy of Flash Continuous Glucose Monitoring (FREESTYLE LIBRE) on the Occurrence of Cardiac Arrhythmias Associated With Hypoglycemia in Patients With Type 2 Diabetes, High Risk of Hypoglycemia and Insulin Therapy : Open-label Randomized Controlled Trial
Brief Title: Efficacy of Flash Glucose-Sensing Technology on the Occurrence of Cardiac Arrhythmias Associated With Hypoglycemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SPIDER-STYLE
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Insulin Treated Type 2 Diabetes With High Risk of Hypoglycemia
Keywords: Freestyle libre; Type 2 diabetes; Hypoglycemia-induced cardiac arrhythmias; Flash Continuous Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flash continuous glucose monitoring system (Experimental): Participants will wear the FREESTYLE LIBRE device and receive a specific therapeutic education for its use.
  Interventions: Device: FREESTYLE LIBRE device, a Flash Continuous Glucose Monitoring System
- Standard self monitoring blood glucose system (Active Comparator): Participants will use their own usual self monitoring blood glucose system and receive a C They will wear a masked FREESTYLE LIBRE Pro system.
  Interventions: Device: Usual self monitoring Blood Glucose device

INTERVENTIONS:
Device: FREESTYLE LIBRE device, a Flash Continuous Glucose Monitoring System — Specific therapeutic education for diabetes self management
  Arms: Flash continuous glucose monitoring system
Device: Usual self monitoring Blood Glucose device — Standard therapeutic education for diabetes self management
  Arms: Standard self monitoring blood glucose system

SUMMARY:
Hypoglycemia, frequently asymptomatic, may lead to cardiac arrythmias and induce an increased risk of cardiovascular morbidity and mortality in patients with type 2 diabetes (T2D). The study hypothesize is that the hypoglycemia reduction, achieved with the FREESTYLE LIBRE device, a Glucose Continuous Monitoring system, may decrease cardiac arrythmias associated with hypoglycemia. So the main objective is to evaluate the efficacy of the FREESTYLE LIBRE system, associated with a specific therapeutic education on the cardiac arrythmias reduction, compared to a capillary ASG system with standard therapeutic education, in patient with T2D with high risk of hypoglycemia.

This is a open, multicenter, controlled, randomized study in parallel group.

ELIGIBILITY:
Inclusion criteria:

* Type 2 diabetes (diagnosis based on the World Health Organization criteria)
* Treatment with insulin therapy (continuous subcutaneous insulin Infusion or more than 1 daily injection)
* Resting heart beat ≥ 60bpm
* High risk of hypoglycemia defined as :

  * Estimated glomerular filtration rate 15-59 ml/min/1.73 m² (according to CKD-EPI formula)
  * Or history of stable proliferative diabetic retinopathy
  * Or body mass index ≤ 30 kg/m²
  * Or history of severe hypoglycemia in the previous 6 months
  * Or history of non-severe ≤70mg/dL hypoglycemia in the previous 4 weeks

Exclusion criteria:

* Type 1 diabetes mellitus or diabetes due to other cause
* History of atrial fibrillation
* Pacemaker
* Estimated glomerular filtration rate <15 ml/min/1.73 m² (according to CKD-EPI formula)
* Currently using a flash continuous Glucose Monitoring device
* In the investigator's opinion, acute or chronic medical condition considered as unsuitable for inclusion in the study .

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-06-29 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of cardiac arrythmic events during a 14 days Continuous ECG Monitoring | 14 days
  Cardiac arrythmic events :
  * Bradycardia < 45 bpm for ≥ 10 seconds
  * or Asystole ≥ 3 seconds
  * or Atrial Fibrillation ≥ 30 seconds
  * or Non-sustained ventricular tachycardia defined as runs of beats arising from the ventricles with duration between 3 beats and 30 s with QRS ≥ 120ms and with RR intervall ≤ 600 ms (>100 bpm)

SECONDARY OUTCOMES:
Prevalence of each component of the primary outcome | 14 days
Prevalence of ≥ 5 minutes Atrial Fibrillation episodes | 14 days
Mean QT interval | First 24 hours
Prevalence of ventricular extrasystoles | First 24 hours

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - University Hospital, Bordeaux, Bordeaux
  - University Hospital, Limoges, Limoges
  - University Hospital, Nantes, Nantes
  - Hospital, Niort, Niort
  - Hospital, Pau, Pau
  - University Hospital, Poitiers, Poitiers
  - University Hospital, Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided